CLINICAL TRIAL: NCT06899022
Title: Investigating the Role of Attention in Perceptual and Cognitive Consequences of Parkinson's Disease
Brief Title: Attention and Eye Movement in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0082-25-FB; P20GM130447 (NIH)
Record Dates: First submitted 2025-03-14; First posted 2025-03-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-03

CONDITIONS: Essential Tremor; Parkinson's Disease (PD)
Keywords: Deep Brain Stimulation; Attention; Perception; Eye movement
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: The interventional component of the study examines whether and how altered level and frequency of deep brain stimulation (DBS) acutely affects eye movement and perception of facial emotion. Participants will be tested in 3 stimulation conditions in random order: normal therapeutic DBS, reduced (50%) current DBS at the normal therapeutic frequency and reduced frequency (4 Hz) at the normal therapeutic current.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute alteration of DBS (Experimental): All participants in the single arm of this study will undergo acute alteration of DBS stimulation under three conditions in randomized order over the course of 1 hour.
  Interventions: Other: Normal therapeutic DBS; Other: Reduced current DBS; Other: Reduced frequency DBS

INTERVENTIONS:
Other: Normal therapeutic DBS — Participants will receive deep brain stimulation delivered at the clinically determined therapeutic frequency and current over approximately 20 min.
Other: Reduced current DBS — Participants will receive deep brain stimulation delivered at the clinically determined therapeutic frequency and reduced (50%) current over approximately 20 minutes.
Other: Reduced frequency DBS — Participants will receive deep brain stimulation delivered at the clinically determined therapeutic current and reduced (4 Hz) frequency over approximately 20 min.

SUMMARY:
The goal of this observational and interventional study is to understand how therapeutic deep brain stimulation (DBS) affects attention, perception and cognition in participants with Parkinson's disease (PD) and essential tremor (ET). The main questions it aims to answer are:

* Does impaired control of attention and eye movement in PD alter how social cues are perceived and interpreted?
* Does therapeutic DBS improve or worsen attentional and perceptual deficits for social cues in PD and ET?
* Can DBS be optimized to restore normal attentional control in PD while remaining an effective therapy for other aspects of the disorder.
* What do parts of the brain targeted by DBS contribute to the control of attention?

Using an eye tracking camera, investigators will study how participants with PD and ET look at and perceive facial expressions of emotion before and after starting DBS therapy, in comparison to a group of healthy participants without ET, PD or DBS. Participants with PD and ET will see and rate morphed facial expressions on a computer screen in three conditions:

* Before starting DBS therapy (over approximately 1 hour).
* In the operating room, during the standard procedure to implant DBS electrodes, while the participant is awake (for no more than 15 minutes).
* After starting DBS therapy, with brief experimental changes of DBS stimulation level and frequency (over approximately 1 hour).

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common age-related neurodegenerative disorder, with approximately 90,000 new cases diagnosed annually in North America. Although motor symptoms define the disorder, PD also leads to cognitive and emotional changes, such as difficulties in recognizing facial expressions and regulating attention, which often overshadow motor issues as the disease progresses. The goal of this study is to better understand the link between attention, eye movement, and emotional perception in PD, testing the hypothesis that disrupted attention leads to altered perception of facial emotions. The study will also investigate how deep brain stimulation (DBS) of the subthalamic nucleus (STN) affects these processes, providing critical insights into the cognitive and perceptual consequences of the treatment.

This research addresses a critical gap in understanding non-motor symptoms of Parkinson's disease by exploring how attention, eye movement, and perception interact. Findings will provide evidence on whether cognitive and emotional symptoms in PD stem from impaired attentional control, offering a new framework for treating these deficits. Additionally, the study will shed light on how different DBS frequencies affect perception and cognition, potentially guiding personalized stimulation strategies to alleviate both motor and non-motor symptoms. The insights gained may influence future therapies for PD, advancing both scientific knowledge and patient care.

Participants will be divided into three groups: PD undergoing DBS, essential tremor (ET) undergoing DBS (as a comparison group for non-PD DBS effects) and healthy age- and sex-matched controls. Participants will complete facial morph rating tasks (rating faces as happy, neutral, or sad) and visual search tasks (finding faces among distractors), while their eye movements are tracked.

The first study aim is to measure how altered attention influences facial emotion perception in PD by tracking eye movements while participants view and categorize emotional face stimuli. The second aim is to characterize brain activity in the STN related to attentional and perceptual processes during awake DBS surgery by capturing microelectrode recordings (MER) of neural activity while participants view emotional faces, allowing researchers to map STN's role in guiding attention and eye movements. The third aim is to test how DBS stimulation at different frequencies (high, low, or off) affects attention, eye movement, and emotional perception by having participants perform visual and perceptual tasks under varying DBS settings to evaluate how brain stimulation influences cognitive and perceptual functions.

ELIGIBILITY:
Inclusion Criteria

* All Participants (Aim 1):

  * Ability and willingness to provide signed informed consent for this study
  * Ability to express perceptual judgments through a button press or mouse- controlled computerized slider
  * Age 19 - 90 years
* DBS Participants (Aim 1):

  * Diagnosis of idiopathic Parkinson's disease (PD) or essential tremor (ET)
  * Scheduled for new implantation of a therapeutic DBS device targeted to subthalamic nucleus (STN), ventral intermediate nucleus of thalamus (VIM) or internal globus pallidus (GPi)
* Comparison Participants (Aim 1):

  o Selection by age matching to participants in PD group
* Parkinson's disease (PD) and essential tremor (ET) Participants (Aim 2):

  * Ability and willingness to provide signed informed consent for this study
  * Ability to express perceptual judgments through a button press or mouse- controlled computerized slider
  * Age 19 - 90 years
  * Scheduled for awake DBS implantation with clinical micro-electrode recordings (MER)
  * Willing and able to engage in tasks during an awake surgical procedure
* Parkinson's disease (PD) and essential tremor (ET) Participants (Aim 3):

  * Ability and willingness to provide signed informed consent for this study
  * Ability to express perceptual judgments through a button press or mouse- controlled computerized slider
  * Age 19 - 90 years
  * Willing to undergo acute manipulations of DBS
  * Able to tolerate acute changes of DBS

Exclusion Criteria

* All Participants (Aim 1):

  * Corrected visual acuity insufficient to perceptually judge face stimuli
  * Inability to understand task instructions or complete task requirements
* DBS Participants (Aim 1):

  o Insufficient therapeutic control of motor symptoms to engage in tasks requiring button press or use of a mouse to control a slider
* Healthy Comparison Participants (Aim 1):

  o History of neurodegenerative disorder
* Parkinson's disease (PD) and essential tremor (ET) Participants (Aim 2):

  * Corrected visual acuity insufficient to perceptually judge face stimuli
  * Inability to understand task instructions or complete task requirements
  * Not undergoing awake DBS implantation
  * Uncorrected visual acuity insufficient to perceptually judge face stimuli
* Parkinson's disease (PD) and essential tremor (ET) Participants (Aim 3):

  * Corrected visual acuity insufficient to perceptually judge face stimuli
  * Inability to understand task instructions or complete task requirements
  * Failure of DBS to achieve a therapeutic effect on motor symptoms

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Facial Expression Rating | Over two experimental sessions, once prior to DBS surgery and once 2-3 weeks after surgery, following clinical optimization of DBS.
  Participants will rate facial expression along a continuous scale using a computerized slider, following the affective bias task (ABT) of Bijanki et al. (2014). The scale is anchored with three descriptors, "Very Sad" at slider value 0 (left), "Neutral", at position 0.5 (middle), and "Very Happy" at 1.0 (right). Responses are compared between two time points: (1) at the initial pre-surgical testing session and post DBS implantation and (2) at the post-implantation session following clinical optimization of therapeutic parameters, 2-3 weeks after surgery. The comparison will examine both the direction of any bias of the rating, against normative ratings, and the magnitude of average deviation from normative ratings. Finally, the ratings will be incorporated into a generalized linear model of gaze position (Kovach 2014) to identify the association between perceived facial expression and characteristic fixation patterns.
Eye Tracking | Over two experimental sessions, once prior to DBS surgery and once 2-3 weeks after surgery, following clinical optimization of DBS.
  The location and duration of gaze fixations will be recorded with a remote eye tracking camera. The location of gaze fixations will be treated as the dependent measure within a generalized linear modeling (GLM) framework for spatial point processes, described in Kovach and Adolphs (2014). Parameter estimates of the model give the log relative risk of fixation at different locations in the visual scene as a function of the independent measures of the model. Independent measures include the main effect of (1) Fourier basis functions encoding scene location and its interactions with (2) image rating in the affective bias task of Bijanki et. al (2014), (3) session and (4) DBS stimulation state. Measures derived from the GLM model will also include the statistical deviation (e.g. Kullback-Leibler divergence) from the average distribution of fixations observed in healthy comparison subjects for each image.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher K Kovach, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McIntyre CC, Hahn PJ. Network perspectives on the mechanisms of deep brain stimulation. Neurobiol Dis. 2010 Jun;38(3):329-37. doi: 10.1016/j.nbd.2009.09.022. Epub 2009 Oct 3. PMID 19804831
- [Background] Sugita Y. Face perception in monkeys reared with no exposure to faces. Proc Natl Acad Sci U S A. 2008 Jan 8;105(1):394-8. doi: 10.1073/pnas.0706079105. Epub 2008 Jan 2. PMID 18172214
- [Background] W. Penny and A. Holmes. Random effects analysis. Statistical parametric mapping: The analysis of functional brain images, 156:165, 2007.
- [Background] C. K. Kovach and M. A. Howard III. Decomposition of higher-order spectra for blind multiple-input deconvolution, pattern identification and separation. Signal Processing, 165:357-379, 2019.
- [Background] C. Kovach, J. Moreira, J. Berger, M. Howard III, L. Gwilliams, A. Fallah, L. Comstock, and E. Mendes. Higher-order spectral decomposition applied to spike sorting. Feb. 2023.
- [Background] Tottenham N, Tanaka JW, Leon AC, McCarry T, Nurse M, Hare TA, Marcus DJ, Westerlund A, Casey BJ, Nelson C. The NimStim set of facial expressions: judgments from untrained research participants. Psychiatry Res. 2009 Aug 15;168(3):242-9. doi: 10.1016/j.psychres.2008.05.006. Epub 2009 Jun 28. PMID 19564050
- [Background] X. Fan, M. Mocchi, B. Pascuzzi, J. Xiao, B. A. Metzger, R. K. Mathura, C. Hacker, J. A. Adkinson, E. Bartoli, S. Elhassa, et al. Brain mechanisms underlying the emotion processing bias in treatment- resistant depression. Nature Mental Health, pages 1-10, 2024.
- [Background] Metzger BA, Kalva P, Mocchi MM, Cui B, Adkinson JA, Wang Z, Mathura R, Kanja K, Gavvala J, Krishnan V, Lin L, Maheshwari A, Shofty B, Magnotti JF, Willie JT, Sheth SA, Bijanki KR. Intracranial stimulation and EEG feature analysis reveal affective salience network specialization. Brain. 2023 Oct 3;146(10):4366-4377. doi: 10.1093/brain/awad200. PMID 37293814
- [Background] Bijanki KR, Kovach CK, McCormick LM, Kawasaki H, Dlouhy BJ, Feinstein J, Jones RD, Howard MA 3rd. Case report: stimulation of the right amygdala induces transient changes in affective bias. Brain Stimul. 2014 Sep-Oct;7(5):690-3. doi: 10.1016/j.brs.2014.05.005. Epub 2014 May 24. PMID 24972588
- [Background] Marneweck M, Loftus A, Hammond G. Psychophysical measures of sensitivity to facial expression of emotion. Front Psychol. 2013 Feb 20;4:63. doi: 10.3389/fpsyg.2013.00063. eCollection 2013. PMID 23431121
- [Background] Sprengelmeyer R, Young AW, Mahn K, Schroeder U, Woitalla D, Buttner T, Kuhn W, Przuntek H. Facial expression recognition in people with medicated and unmedicated Parkinson's disease. Neuropsychologia. 2003;41(8):1047-57. doi: 10.1016/s0028-3932(02)00295-6. PMID 12667540
- [Background] Hershey T, Campbell MC, Videen TO, Lugar HM, Weaver PM, Hartlein J, Karimi M, Tabbal SD, Perlmutter JS. Mapping Go-No-Go performance within the subthalamic nucleus region. Brain. 2010 Dec;133(Pt 12):3625-34. doi: 10.1093/brain/awq256. Epub 2010 Sep 20. PMID 20855421
- [Background] McIntosh LG, Mannava S, Camalier CR, Folley BS, Albritton A, Konrad PE, Charles D, Park S, Neimat JS. Emotion recognition in early Parkinson's disease patients undergoing deep brain stimulation or dopaminergic therapy: a comparison to healthy participants. Front Aging Neurosci. 2015 Jan 21;6:349. doi: 10.3389/fnagi.2014.00349. eCollection 2014. PMID 25653616
- [Background] Albuquerque L, Coelho M, Martins M, Guedes LC, Rosa MM, Ferreira JJ, Cattoni MB, Carvalho H, Ferreira AG, Martins IP. STN-DBS does not change emotion recognition in advanced Parkinson's disease. Parkinsonism Relat Disord. 2014 Feb;20(2):166-9. doi: 10.1016/j.parkreldis.2013.10.010. Epub 2013 Oct 18. PMID 24182523
- [Background] Berney A, Panisset M, Sadikot AF, Ptito A, Dagher A, Fraraccio M, Savard G, Pell M, Benkelfat C. Mood stability during acute stimulator challenge in Parkinson's disease patients under long-term treatment with subthalamic deep brain stimulation. Mov Disord. 2007 Jun 15;22(8):1093-6. doi: 10.1002/mds.21245. PMID 17394245
- [Background] Schneider F, Habel U, Volkmann J, Regel S, Kornischka J, Sturm V, Freund HJ. Deep brain stimulation of the subthalamic nucleus enhances emotional processing in Parkinson disease. Arch Gen Psychiatry. 2003 Mar;60(3):296-302. doi: 10.1001/archpsyc.60.3.296. PMID 12622663
- [Background] Wagenbreth C, Wattenberg L, Heinze HJ, Zaehle T. Implicit and explicit processing of emotional facial expressions in Parkinson's disease. Behav Brain Res. 2016 Apr 15;303:182-90. doi: 10.1016/j.bbr.2016.01.059. Epub 2016 Feb 2. PMID 26850933
- [Background] Mermillod M, Mondillon L, Rieu I, Devaux D, Chambres P, Auxiette C, Dalens H, Coulangeon LM, Jalenques I, Durif F. Dopamine replacement therapy and deep brain stimulation of the subthalamic nuclei induce modulation of emotional processes at different spatial frequencies in Parkinson's disease. J Parkinsons Dis. 2014;4(1):97-110. doi: 10.3233/JPD-130256. PMID 24496100
- [Background] Mondillon L, Mermillod M, Musca SC, Rieu I, Vidal T, Chambres P, Auxiette C, Dalens H, Marie Coulangeon L, Jalenques I, Lemaire JJ, Ulla M, Derost P, Marques A, Durif F. The combined effect of subthalamic nuclei deep brain stimulation and L-dopa increases emotion recognition in Parkinson's disease. Neuropsychologia. 2012 Oct;50(12):2869-2879. doi: 10.1016/j.neuropsychologia.2012.08.016. Epub 2012 Aug 28. PMID 22944002
- [Background] Peron J, Biseul I, Leray E, Vicente S, Le Jeune F, Drapier S, Drapier D, Sauleau P, Haegelen C, Verin M. Subthalamic nucleus stimulation affects fear and sadness recognition in Parkinson's disease. Neuropsychology. 2010 Jan;24(1):1-8. doi: 10.1037/a0017433. PMID 20063943
- [Background] Drapier D, Peron J, Leray E, Sauleau P, Biseul I, Drapier S, Le Jeune F, Travers D, Bourguignon A, Haegelen C, Millet B, Verin M. Emotion recognition impairment and apathy after subthalamic nucleus stimulation in Parkinson's disease have separate neural substrates. Neuropsychologia. 2008 Sep;46(11):2796-801. doi: 10.1016/j.neuropsychologia.2008.05.006. Epub 2008 May 20. PMID 18579165
- [Background] Biseul I, Sauleau P, Haegelen C, Trebon P, Drapier D, Raoul S, Drapier S, Lallement F, Rivier I, Lajat Y, Verin M. Fear recognition is impaired by subthalamic nucleus stimulation in Parkinson's disease. Neuropsychologia. 2005;43(7):1054-9. doi: 10.1016/j.neuropsychologia.2004.10.006. Epub 2004 Dec 30. PMID 15769491
- [Background] Dujardin K, Blairy S, Defebvre L, Krystkowiak P, Hess U, Blond S, Destee A. Subthalamic nucleus stimulation induces deficits in decoding emotional facial expressions in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2004 Feb;75(2):202-8. PMID 14742588
- [Background] Schroeder U, Kuehler A, Hennenlotter A, Haslinger B, Tronnier VM, Krause M, Pfister R, Sprengelmeyer R, Lange KW, Ceballos-Baumann AO. Facial expression recognition and subthalamic nucleus stimulation. J Neurol Neurosurg Psychiatry. 2004 Apr;75(4):648-50. doi: 10.1136/jnnp.2003.019794. PMID 15026519
- [Background] Pinkhardt EH, Jurgens R, Lule D, Heimrath J, Ludolph AC, Becker W, Kassubek J. Eye movement impairments in Parkinson's disease: possible role of extradopaminergic mechanisms. BMC Neurol. 2012 Feb 29;12:5. doi: 10.1186/1471-2377-12-5. PMID 22375860
- [Background] Dec-Cwiek M, Tutaj M, Gracies JM, Volkmann J, Rudzinska M, Slowik A, Szczudlik A. Opposite effects of l-dopa and DBS-STN on saccadic eye movements in advanced Parkinson's disease. Neurol Neurochir Pol. 2017 Sep-Oct;51(5):354-360. doi: 10.1016/j.pjnns.2017.06.002. Epub 2017 Jun 24. PMID 28669542
- [Background] Temel Y, Visser-Vandewalle V, Carpenter RHS. Saccadic latency during electrical stimulation of the human subthalamic nucleus. Curr Biol. 2008 May 20;18(10):R412-R414. doi: 10.1016/j.cub.2008.03.008. No abstract available. PMID 18492468
- [Background] Fischer P, Ossandon JP, Keyser J, Gulberti A, Wilming N, Hamel W, Koppen J, Buhmann C, Westphal M, Gerloff C, Moll CK, Engel AK, Konig P. STN-DBS Reduces Saccadic Hypometria but Not Visuospatial Bias in Parkinson's Disease Patients. Front Behav Neurosci. 2016 May 3;10:85. doi: 10.3389/fnbeh.2016.00085. eCollection 2016. PMID 27199693
- [Background] Nilsson MH, Patel M, Rehncrona S, Magnusson M, Fransson PA. Subthalamic deep brain stimulation improves smooth pursuit and saccade performance in patients with Parkinson's disease. J Neuroeng Rehabil. 2013 Apr 3;10:33. doi: 10.1186/1743-0003-10-33. PMID 23551890
- [Background] Klarendic M, Kaski D. Deep brain stimulation and eye movements. Eur J Neurosci. 2021 Apr;53(7):2344-2361. doi: 10.1111/ejn.14898. Epub 2020 Jul 27. PMID 32643303
- [Background] Fawcett AP, Cunic D, Hamani C, Hodaie M, Lozano AM, Chen R, Hutchison WD. Saccade-related potentials recorded from human subthalamic nucleus. Clin Neurophysiol. 2007 Jan;118(1):155-63. doi: 10.1016/j.clinph.2006.09.016. Epub 2006 Nov 9. PMID 17097341
- [Background] Kovach CK, Adolphs R. Investigating attention in complex visual search. Vision Res. 2015 Nov;116(Pt B):127-41. doi: 10.1016/j.visres.2014.11.011. Epub 2014 Dec 8. PMID 25499190
- [Background] Kovach CK, Sutterer MJ, Rushia SN, Teriakidis A, Jenison RL. Two systems drive attention to rewards. Front Psychol. 2014 Feb 5;5:46. doi: 10.3389/fpsyg.2014.00046. eCollection 2014. PMID 24550868
- [Background] Beylergil SB, Kilbane C, Shaikh AG, Ghasia FF. Eye movements in Parkinson's disease during visual search. J Neurol Sci. 2022 Sep 15;440:120299. doi: 10.1016/j.jns.2022.120299. Epub 2022 May 28. PMID 35810513
- [Background] Waldthaler J, Stock L, Student J, Sommerkorn J, Dowiasch S, Timmermann L. Antisaccades in Parkinson's Disease: A Meta-Analysis. Neuropsychol Rev. 2021 Dec;31(4):628-642. doi: 10.1007/s11065-021-09489-1. Epub 2021 Mar 19. PMID 33742354
- [Background] Clark US, Neargarder S, Cronin-Golomb A. Visual exploration of emotional facial expressions in Parkinson's disease. Neuropsychologia. 2010 Jun;48(7):1901-13. doi: 10.1016/j.neuropsychologia.2010.03.006. Epub 2010 Mar 15. PMID 20230847
- [Background] Hodgson TL, Tiesman B, Owen AM, Kennard C. Abnormal gaze strategies during problem solving in Parkinson's disease. Neuropsychologia. 2002;40(4):411-22. doi: 10.1016/s0028-3932(01)00099-9. PMID 11684174
- [Background] Antoniades CA, Spering M. Eye movements in Parkinson's disease: from neurophysiological mechanisms to diagnostic tools. Trends Neurosci. 2024 Jan;47(1):71-83. doi: 10.1016/j.tins.2023.11.001. Epub 2023 Dec 2. PMID 38042680
- [Background] Zhang Y, Yan A, Liu B, Wan Y, Zhao Y, Liu Y, Tan J, Song L, Gu Y, Liu Z. Oculomotor Performances Are Associated With Motor and Non-motor Symptoms in Parkinson's Disease. Front Neurol. 2018 Nov 28;9:960. doi: 10.3389/fneur.2018.00960. eCollection 2018. PMID 30546341
- [Background] Pretegiani E, Optican LM. Eye Movements in Parkinson's Disease and Inherited Parkinsonian Syndromes. Front Neurol. 2017 Nov 9;8:592. doi: 10.3389/fneur.2017.00592. eCollection 2017. PMID 29170650
- [Background] Pinkhardt EH, Kassubek J. Ocular motor abnormalities in Parkinsonian syndromes. Parkinsonism Relat Disord. 2011 May;17(4):223-30. doi: 10.1016/j.parkreldis.2010.08.004. Epub 2010 Aug 30. PMID 20801069
- [Background] Shibasaki H, Tsuji S, Kuroiwa Y. Oculomotor abnormalities in Parkinson's disease. Arch Neurol. 1979 Jun;36(6):360-4. doi: 10.1001/archneur.1979.00500420070009. PMID 454234
- [Background] Assogna F, Pontieri FE, Caltagirone C, Spalletta G. The recognition of facial emotion expressions in Parkinson's disease. Eur Neuropsychopharmacol. 2008 Nov;18(11):835-48. doi: 10.1016/j.euroneuro.2008.07.004. Epub 2008 Aug 15. PMID 18707851
- [Background] Pell MD, Leonard CL. Facial expression decoding in early Parkinson's disease. Brain Res Cogn Brain Res. 2005 May;23(2-3):327-40. doi: 10.1016/j.cogbrainres.2004.11.004. Epub 2005 Jan 7. PMID 15820640
- [Background] Adolphs R, Schul R, Tranel D. Intact recognition of facial emotion in Parkinson's disease. Neuropsychology. 1998 Apr;12(2):253-8. doi: 10.1037//0894-4105.12.2.253. PMID 9556771
- [Background] Dodich A, Funghi G, Meli C, Pennacchio M, Longo C, Malaguti MC, Di Giacopo R, Zappini F, Turella L, Papagno C. Deficits in Emotion Recognition and Theory of Mind in Parkinson's Disease Patients With and Without Cognitive Impairments. Front Psychol. 2022 May 13;13:866809. doi: 10.3389/fpsyg.2022.866809. eCollection 2022. PMID 35645902
- [Background] Mattavelli G, Barvas E, Longo C, Zappini F, Ottaviani D, Malaguti MC, Pellegrini M, Papagno C. Facial expressions recognition and discrimination in Parkinson's disease. J Neuropsychol. 2021 Mar;15(1):46-68. doi: 10.1111/jnp.12209. Epub 2020 Apr 22. PMID 32319735
- [Background] Coundouris SP, Adams AG, Grainger SA, Henry JD. Social perceptual function in parkinson's disease: A meta-analysis. Neurosci Biobehav Rev. 2019 Sep;104:255-267. doi: 10.1016/j.neubiorev.2019.07.011. Epub 2019 Jul 20. PMID 31336113
- [Background] Marneweck M, Hammond G. Discriminating facial expressions of emotion and its link with perceiving visual form in Parkinson's disease. J Neurol Sci. 2014 Nov 15;346(1-2):149-55. doi: 10.1016/j.jns.2014.08.014. Epub 2014 Aug 20. PMID 25179875
- [Background] Ariatti A, Benuzzi F, Nichelli P. Recognition of emotions from visual and prosodic cues in Parkinson's disease. Neurol Sci. 2008 Sep;29(4):219-27. doi: 10.1007/s10072-008-0971-9. Epub 2008 Sep 20. PMID 18810595
- [Background] Suzuki A, Hoshino T, Shigemasu K, Kawamura M. Disgust-specific impairment of facial expression recognition in Parkinson's disease. Brain. 2006 Mar;129(Pt 3):707-17. doi: 10.1093/brain/awl011. Epub 2006 Jan 16. PMID 16415306
- [Background] Dujardin K, Blairy S, Defebvre L, Duhem S, Noel Y, Hess U, Destee A. Deficits in decoding emotional facial expressions in Parkinson's disease. Neuropsychologia. 2004;42(2):239-50. doi: 10.1016/s0028-3932(03)00154-4. PMID 14644109
- [Background] Simons G, Pasqualini MC, Reddy V, Wood J. Emotional and nonemotional facial expressions in people with Parkinson's disease. J Int Neuropsychol Soc. 2004 Jul;10(4):521-35. doi: 10.1017/S135561770410413X. PMID 15327731
- [Background] Prenger MTM, Madray R, Van Hedger K, Anello M, MacDonald PA. Social Symptoms of Parkinson's Disease. Parkinsons Dis. 2020 Dec 31;2020:8846544. doi: 10.1155/2020/8846544. eCollection 2020. PMID 33489081
- [Background] Pell MD, Monetta L, Rothermich K, Kotz SA, Cheang HS, McDonald S. Social perception in adults with Parkinson's disease. Neuropsychology. 2014 Nov;28(6):905-16. doi: 10.1037/neu0000090. Epub 2014 Jun 2. PMID 24885448
- [Background] Peron J, Dondaine T, Le Jeune F, Grandjean D, Verin M. Emotional processing in Parkinson's disease: a systematic review. Mov Disord. 2012 Feb;27(2):186-99. doi: 10.1002/mds.24025. Epub 2011 Dec 9. PMID 22162004
- [Background] Caap-Ahlgren M, Dehlin O. Factors of importance to the caregiver burden experienced by family caregivers of Parkinson's disease patients. Aging Clin Exp Res. 2002 Oct;14(5):371-7. doi: 10.1007/BF03324464. PMID 12602571
- [Background] Jacobs DH, Shuren J, Bowers D, Heilman KM. Emotional facial imagery, perception, and expression in Parkinson's disease. Neurology. 1995 Sep;45(9):1696-702. doi: 10.1212/wnl.45.9.1696. PMID 7675229
- [Background] Isoda M, Hikosaka O. Switching from automatic to controlled action by monkey medial frontal cortex. Nat Neurosci. 2007 Feb;10(2):240-8. doi: 10.1038/nn1830. Epub 2007 Jan 21. PMID 17237780
- [Background] Siegert RJ, Taylor KD, Weatherall M, Abernethy DA. Is implicit sequence learning impaired in Parkinson's disease? A meta-analysis. Neuropsychology. 2006 Jul;20(4):490-5. doi: 10.1037/0894-4105.20.4.490. PMID 16846267
- [Background] Jahanshahi M, Obeso I, Rothwell JC, Obeso JA. A fronto-striato-subthalamic-pallidal network for goal-directed and habitual inhibition. Nat Rev Neurosci. 2015 Dec;16(12):719-32. doi: 10.1038/nrn4038. Epub 2015 Nov 4. PMID 26530468
- [Background] Doyon J, Bellec P, Amsel R, Penhune V, Monchi O, Carrier J, Lehericy S, Benali H. Contributions of the basal ganglia and functionally related brain structures to motor learning. Behav Brain Res. 2009 Apr 12;199(1):61-75. doi: 10.1016/j.bbr.2008.11.012. Epub 2008 Nov 17. PMID 19061920
- [Background] Arcaro MJ, Schade PF, Vincent JL, Ponce CR, Livingstone MS. Seeing faces is necessary for face-domain formation. Nat Neurosci. 2017 Oct;20(10):1404-1412. doi: 10.1038/nn.4635. Epub 2017 Sep 4. PMID 28869581
- [Background] Kundel HL, Nodine CF, Krupinski EA, Mello-Thoms C. Using gaze-tracking data and mixture distribution analysis to support a holistic model for the detection of cancers on mammograms. Acad Radiol. 2008 Jul;15(7):881-6. doi: 10.1016/j.acra.2008.01.023. PMID 18572124
- [Background] Charness N, Reingold EM, Pomplun M, Stampe DM. The perceptual aspect of skilled performance in chess: evidence from eye movements. Mem Cognit. 2001 Dec;29(8):1146-52. doi: 10.3758/bf03206384. PMID 11913751
- [Background] Wolfe JM, Butcher SJ, Lee C, Hyle M. Changing your mind: on the contributions of top-down and bottom-up guidance in visual search for feature singletons. J Exp Psychol Hum Percept Perform. 2003 Apr;29(2):483-502. doi: 10.1037/0096-1523.29.2.483. PMID 12760630
- [Background] Braak H, Del Tredici K. Invited Article: Nervous system pathology in sporadic Parkinson disease. Neurology. 2008 May 13;70(20):1916-25. doi: 10.1212/01.wnl.0000312279.49272.9f. No abstract available. PMID 18474848
- [Background] Brown RG, Marsden CD. Internal versus external cues and the control of attention in Parkinson's disease. Brain. 1988 Apr;111 ( Pt 2):323-45. doi: 10.1093/brain/111.2.323. PMID 3378139
- [Background] Schurgin MW, Nelson J, Iida S, Ohira H, Chiao JY, Franconeri SL. Eye movements during emotion recognition in faces. J Vis. 2014 Nov 18;14(13):14. doi: 10.1167/14.13.14. PMID 25406159
- [Background] Oberauer K. Working Memory and Attention - A Conceptual Analysis and Review. J Cogn. 2019 Aug 8;2(1):36. doi: 10.5334/joc.58. PMID 31517246
- [Background] D. A. Norman and T. Shallice. Attention to action: Willed and automatic control of behavior. In R. Davidson, G. Schwartz, and S. D, editors, Consciousness and self regulation: Advances in Research, Volume IV. New York: Plenum Press, 1986.
- [Background] Dirnberger G, Jahanshahi M. Executive dysfunction in Parkinson's disease: a review. J Neuropsychol. 2013 Sep;7(2):193-224. doi: 10.1111/jnp.12028. PMID 24007368
- [Background] Ho MW, Chien SH, Lu MK, Chen JC, Aoh Y, Chen CM, Lane HY, Tsai CH. Impairments in face discrimination and emotion recognition are related to aging and cognitive dysfunctions in Parkinson's disease with dementia. Sci Rep. 2020 Mar 9;10(1):4367. doi: 10.1038/s41598-020-61310-w. PMID 32152359
- [Background] K. E. Thorpe, A. I. Levey, and J. Thomas. Us burden of neurodegenerative disease. Partnership to Fight Chronic Disease (PFCD), pages 1-13, 2021.
- [Background] Yang W, Hamilton JL, Kopil C, Beck JC, Tanner CM, Albin RL, Ray Dorsey E, Dahodwala N, Cintina I, Hogan P, Thompson T. Current and projected future economic burden of Parkinson's disease in the U.S. NPJ Parkinsons Dis. 2020 Jul 9;6:15. doi: 10.1038/s41531-020-0117-1. eCollection 2020. PMID 32665974
- [Background] Dorsey ER, Sherer T, Okun MS, Bloem BR. The Emerging Evidence of the Parkinson Pandemic. J Parkinsons Dis. 2018;8(s1):S3-S8. doi: 10.3233/JPD-181474. PMID 30584159
- [Background] Willis AW, Roberts E, Beck JC, Fiske B, Ross W, Savica R, Van Den Eeden SK, Tanner CM, Marras C; Parkinson's Foundation P4 Group. Incidence of Parkinson disease in North America. NPJ Parkinsons Dis. 2022 Dec 15;8(1):170. doi: 10.1038/s41531-022-00410-y. PMID 36522332
- [Background] Kelley R, Flouty O, Emmons EB, Kim Y, Kingyon J, Wessel JR, Oya H, Greenlee JD, Narayanan NS. A human prefrontal-subthalamic circuit for cognitive control. Brain. 2018 Jan 1;141(1):205-216. doi: 10.1093/brain/awx300. PMID 29190362
- [Background] Yugeta A, Terao Y, Fukuda H, Hikosaka O, Yokochi F, Okiyama R, Taniguchi M, Takahashi H, Hamada I, Hanajima R, Ugawa Y. Effects of STN stimulation on the initiation and inhibition of saccade in Parkinson disease. Neurology. 2010 Mar 2;74(9):743-8. doi: 10.1212/WNL.0b013e3181d31e0b. PMID 20194913
- [Background] Isoda M, Hikosaka O. Role for subthalamic nucleus neurons in switching from automatic to controlled eye movement. J Neurosci. 2008 Jul 9;28(28):7209-18. doi: 10.1523/JNEUROSCI.0487-08.2008. PMID 18614691
- [Background] Waldthaler J, Kruger-Zechlin C, Stock L, Deeb Z, Timmermann L. New insights into facial emotion recognition in Parkinson's disease with and without mild cognitive impairment from visual scanning patterns. Clin Park Relat Disord. 2019 Nov 20;1:102-108. doi: 10.1016/j.prdoa.2019.11.003. eCollection 2019. PMID 34316611
- [Background] Hannula DE, Althoff RR, Warren DE, Riggs L, Cohen NJ, Ryan JD. Worth a glance: using eye movements to investigate the cognitive neuroscience of memory. Front Hum Neurosci. 2010 Oct 8;4:166. doi: 10.3389/fnhum.2010.00166. eCollection 2010. PMID 21151363
- [Background] Frei K. Abnormalities of smooth pursuit in Parkinson's disease: A systematic review. Clin Park Relat Disord. 2020 Dec 17;4:100085. doi: 10.1016/j.prdoa.2020.100085. eCollection 2021. PMID 34316663
- [Background] de Haan B, Morgan PS, Rorden C. Covert orienting of attention and overt eye movements activate identical brain regions. Brain Res. 2008 Apr 14;1204:102-11. doi: 10.1016/j.brainres.2008.01.105. Epub 2008 Feb 19. PMID 18329633
- [Background] Tokushige SI, Matsuda SI, Oyama G, Shimo Y, Umemura A, Sasaki T, Inomata-Terada S, Yugeta A, Hamada M, Ugawa Y, Tsuji S, Hattori N, Terao Y. Effect of subthalamic nucleus deep brain stimulation on visual scanning. Clin Neurophysiol. 2018 Nov;129(11):2421-2432. doi: 10.1016/j.clinph.2018.08.003. Epub 2018 Aug 30. PMID 30292079
- [Background] Fawcett AP, Gonzalez EG, Moro E, Steinbach MJ, Lozano AM, Hutchison WD. Subthalamic nucleus deep brain stimulation improves saccades in Parkinson's disease. Neuromodulation. 2010 Jan;13(1):17-25. doi: 10.1111/j.1525-1403.2009.00246.x. Epub 2009 Nov 13. PMID 21992760
- [Background] Blekher T, Weaver M, Rupp J, Nichols WC, Hui SL, Gray J, Yee RD, Wojcieszek J, Foroud T. Multiple step pattern as a biomarker in Parkinson disease. Parkinsonism Relat Disord. 2009 Aug;15(7):506-10. doi: 10.1016/j.parkreldis.2009.01.002. Epub 2009 Feb 10. PMID 19211293
- [Background] Hikosaka O, Takikawa Y, Kawagoe R. Role of the basal ganglia in the control of purposive saccadic eye movements. Physiol Rev. 2000 Jul;80(3):953-78. doi: 10.1152/physrev.2000.80.3.953. PMID 10893428
- [Background] Lieberman A. Depression in Parkinson's disease -- a review. Acta Neurol Scand. 2006 Jan;113(1):1-8. doi: 10.1111/j.1600-0404.2006.00536.x. PMID 16367891
- [Background] Bek J, Poliakoff E, Lander K. Measuring emotion recognition by people with Parkinson's disease using eye-tracking with dynamic facial expressions. J Neurosci Methods. 2020 Feb 1;331:108524. doi: 10.1016/j.jneumeth.2019.108524. Epub 2019 Nov 17. PMID 31747554
- [Background] Wagenbreth C, Kuehne M, Heinze HJ, Zaehle T. Deep Brain Stimulation of the Subthalamic Nucleus Influences Facial Emotion Recognition in Patients With Parkinson's Disease: A Review. Front Psychol. 2019 Dec 3;10:2638. doi: 10.3389/fpsyg.2019.02638. eCollection 2019. PMID 31849760
- [Background] Argaud S, Verin M, Sauleau P, Grandjean D. Facial emotion recognition in Parkinson's disease: A review and new hypotheses. Mov Disord. 2018 Apr;33(4):554-567. doi: 10.1002/mds.27305. Epub 2018 Feb 23. PMID 29473661
- [Background] Assogna F, Cravello L, Orfei MD, Cellupica N, Caltagirone C, Spalletta G. Alexithymia in Parkinson's disease: A systematic review of the literature. Parkinsonism Relat Disord. 2016 Jul;28:1-11. doi: 10.1016/j.parkreldis.2016.03.021. Epub 2016 Mar 30. PMID 27086264
- [Background] Gray HM, Tickle-Degnen L. A meta-analysis of performance on emotion recognition tasks in Parkinson's disease. Neuropsychology. 2010 Mar;24(2):176-91. doi: 10.1037/a0018104. PMID 20230112
- [Background] Clark US, Neargarder S, Cronin-Golomb A. Specific impairments in the recognition of emotional facial expressions in Parkinson's disease. Neuropsychologia. 2008;46(9):2300-9. doi: 10.1016/j.neuropsychologia.2008.03.014. Epub 2008 Mar 30. PMID 18485422
- [Background] Yip JT, Lee TM, Ho SL, Tsang KL, Li LS. Emotion recognition in patients with idiopathic Parkinson's disease. Mov Disord. 2003 Oct;18(10):1115-22. doi: 10.1002/mds.10497. PMID 14534914
- [Background] Soh C, Hervault M, Chalkley NH, Moore CM, Rohl A, Zhang Q, Uc EY, Greenlee JDW, Wessel JR. The human subthalamic nucleus transiently inhibits active attentional processes. Brain. 2024 Sep 3;147(9):3204-3215. doi: 10.1093/brain/awae068. PMID 38436939
- [Background] Lawson RA, Yarnall AJ, Duncan GW, Breen DP, Khoo TK, Williams-Gray CH, Barker RA, Collerton D, Taylor JP, Burn DJ; ICICLE-PD study group. Cognitive decline and quality of life in incident Parkinson's disease: The role of attention. Parkinsonism Relat Disord. 2016 Jun;27:47-53. doi: 10.1016/j.parkreldis.2016.04.009. Epub 2016 Apr 11. PMID 27094482
- [Background] Botha H, Carr J. Attention and visual dysfunction in Parkinson's disease. Parkinsonism Relat Disord. 2012 Jul;18(6):742-7. doi: 10.1016/j.parkreldis.2012.03.004. Epub 2012 Apr 11. PMID 22503538
- [Background] Stam CJ, Visser SL, Op de Coul AA, De Sonneville LM, Schellens RL, Brunia CH, de Smet JS, Gielen G. Disturbed frontal regulation of attention in Parkinson's disease. Brain. 1993 Oct;116 ( Pt 5):1139-58. doi: 10.1093/brain/116.5.1139. PMID 8221052
- [Background] Wright MJ, Burns RJ, Geffen GM, Geffen LB. Covert orientation of visual attention in Parkinson's disease: an impairment in the maintenance of attention. Neuropsychologia. 1990;28(2):151-9. doi: 10.1016/0028-3932(90)90097-8. PMID 2314570
- [Background] LeWitt PA, Chaudhuri KR. Unmet needs in Parkinson disease: Motor and non-motor. Parkinsonism Relat Disord. 2020 Nov;80 Suppl 1:S7-S12. doi: 10.1016/j.parkreldis.2020.09.024. Epub 2020 Dec 19. PMID 33349582
- [Background] Goldman JG, Vernaleo BA, Camicioli R, Dahodwala N, Dobkin RD, Ellis T, Galvin JE, Marras C, Edwards J, Fields J, Golden R, Karlawish J, Levin B, Shulman L, Smith G, Tangney C, Thomas CA, Troster AI, Uc EY, Coyan N, Ellman C, Ellman M, Hoffman C, Hoffman S, Simmonds D. Cognitive impairment in Parkinson's disease: a report from a multidisciplinary symposium on unmet needs and future directions to maintain cognitive health. NPJ Parkinsons Dis. 2018 Jun 26;4:19. doi: 10.1038/s41531-018-0055-3. eCollection 2018. PMID 29951580
- [Background] Dubois B, Pillon B. Cognitive deficits in Parkinson's disease. J Neurol. 1997 Jan;244(1):2-8. doi: 10.1007/pl00007725. PMID 9007738